CLINICAL TRIAL: NCT03404661
Title: Optical and Biochemical Biomarkers in Early Pancreatic Cancer Significance: A Prospective Study
Brief Title: Optical and Biochemical Biomarkers in Early Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Massimo Raimondo, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 17-005211
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Secretin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20cc of venous blood In case of pancreatic cyst, excess fluid above 2cc Excess tumor tissue including portions of cancer and normal tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Pancreas Cancer Subjects: Patients with pancreas cancer will receive Synthetic Human Secretin during an endoscopy procedure.
  Interventions: Drug: Synthetic Human Secretin
- Control Subjects: Controls will receive Synthetic Human Secretin during an endoscopy procedure. Controls are at an elevated risk of pancreas cancer, including pancreatic cystic neoplasms.
  Interventions: Drug: Synthetic Human Secretin
- Familial Pancreatic Cancer Subjects: Subjects who have a family history of pancreas cancer will receive Synthetic Human Secretin during an endoscopy procedure.
  Interventions: Drug: Synthetic Human Secretin

INTERVENTIONS:
Drug: Synthetic Human Secretin — Subjects will receive a dose of 0.2ng/kg while the endoscope is positioned in the second portion of the duodenum.
  Other Names: ChiRhoStim

SUMMARY:
The purpose of this study is to develop a test for detection of pancreatic cancer by looking at the subject's DNA.

DETAILED DESCRIPTION:
Pancreatic juice collection is performed by intravenous injection of FDA approved synthetic human secretin (ChiRhoClin Inc., Burtonsville, MD) at a dose of 0.2 µg/kg will be administered while the endoscope is positioned in the second portion of the duodenum. From within the duodenum and without cannulation of the papilla of Vater, a 2.3-mm plastic aspiration catheter (Olympus, Tokyo, Japan) will be passed through the biopsy channel of the endoscope until visible on screen in the endoscopic monitor. Once active visible secretion via the papilla has begun, the first 10 ml of pancreatic juice will be collected via suctioning. This entire process from secretin injection to sample collection takes an average of 5 minutes. The sample is then aliquoted into 2 ml ampules, which are snap-frozen in liquid nitrogen (or portable rapid-freeze freezer) and freezer-stored until the assays are performed. The top 10 candidate markers from discovery and validation on tissue (AUCs >0.95) and from pilot pancreatic-juice testing (AUCs >0.9) will be evaluated in this study. Following extraction from an equivalent of 0.4 ml pancreatic juice, DNA will be bisulfite treated using optimized methods. Then, an assay of aberrant methylation on target genes will be conducted using the QuARTS technique. Results will be normalized to either a human DNA marker (eg, beta-actin) or a methylated DNA marker identified for normal pancreatic epithelium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred for the evaluation of pancreas cancer, pancreatic cystic neoplasm, and family history of pancreas cancer.
* International normalized ratio (INR) less than 1.5
* Platelet count >50,000

Exclusion Criteria:

* Any medical condition that preclude the patient from having a therapeutic procedure regardless of the Endoscopic ultrasound (EUS) finding
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreas cancer, controls at an elevated risk of pancreas cancer, including pancreatic cystic neoplasms, and subjects with a familial history of pancreas cancer.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Methylated DNA markers as measured by mean percentage of total human DNA per pancreatic juice volume | one year
  After pancreatic juice is collected, top 10 markers for pancreas cancer detection will be done from discovery and validation on tissue (AUC>.95) and from pilot pancreatic-juice testing (AUCs >0.9).

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Raimondo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials